CLINICAL TRIAL: NCT00827840
Title: Paliperidone ER Versus Risperidone for Neurocognitive Function in Patients With Schizophrenia: a Randomized, Open-label, Controlled Trial
Brief Title: Paliperidone Extended-Release (ER) Versus Risperidone for Neurocognitive Function in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry); Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jin-Sang Yoon, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAL-KOR-9006
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Paliperidone ER (Experimental): New antipsychotics
  Interventions: Drug: Paliperidone ER
- 2 Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Paliperidone ER — 3mg to 12mg of Paliperidone ER once a day
  Other Names: Invega
  Arms: 1. Paliperidone ER
Drug: Risperidone — 1 to 6 mg of risperidone once or twice a day
  Other Names: Risperdal
  Arms: 2 Risperidone

SUMMARY:
Primary objective: To examine whether the switch to paliperidone ER from risperidone improves cognitive function in stabilized patients with schizophrenia.

Secondary objectives: To compare the general clinical outcomes (efficacy and safety) after switching to paliperidone ER from risperidone

DETAILED DESCRIPTION:
This is a 12-week, randomized, parallel-group, open labeled, flexible-dose study. The patients will be randomized to the risperidone-continuation group in which they continue to receive risperidone, or to the paliperidone-switch group in which they are switched from risperidone to paliperidone. In the paliperidone-switch group, risperidone will be tapered off during the first 4 weeks of the study, while paliperidone is titrated simultaneously. The doses of both drugs will be adjusted according to the clinical judgment of each research psychiatrist, within 6 mg/day of risperidone and 12 mg/day of paliperidone.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as schizophrenia by DSM-IV-TR criteria both in inpatients
* Patients who are symptomatically stable, as judged by the treating psychiatrist, and receive a stable dose of risperidone for a minimum of 2 weeks before enrollment.
* Patients with ability to complete various questionnaires.
* Patients and/or their legal guardians/representatives who sufficiently understand the objective of the study and sign informed consent form

Exclusion Criteria:

* Active psychotic symptoms, including severe behavioral disturbance
* Relevant history of or current presence of any significant or unstable medical disease
* A woman who is pregnant, breast-feeding or planning to become pregnant during the study period
* Patients with the history of serious allergy or multiple adverse drug reactions
* Patients with the history of taking paliperidone ER within 60 days
* Patients with history of taking clozapine within 60 days
* Patients who require the treatment of other medications influencing CNS, except permitted concomitant drugs in advance

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Neurocognitive function | 12 weeks

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Sang Yoon, Professor, Principal Investigator — Dept. of Psychiatry, Chonnam National University Hospital
Locations (1):
- Dept. of Psychiatry, Chonnam National Univeristy Hospital, Gwangju, South Korea

REFERENCES:
- [Derived] Kim SW, Chung YC, Lee YH, Lee JH, Kim SY, Bae KY, Kim JM, Shin IS, Yoon JS. Paliperidone ER versus risperidone for neurocognitive function in patients with schizophrenia: a randomized, open-label, controlled trial. Int Clin Psychopharmacol. 2012 Sep;27(5):267-74. doi: 10.1097/YIC.0b013e328356acad. PMID 22809972